CLINICAL TRIAL: NCT05223634
Title: A Semi-Quantitative and Comparative Study for the Detection of Group A β-Hemolytic Streptococci in Oral Samples
Brief Title: Detection of Group A β-Hemolytic Streptococci in Oral Samples
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hero Scientific (Industry)
Responsible Party: Sponsor
Other Study IDs: STRP.P002
Record Dates: First submitted 2022-01-03; First posted 2022-02-04 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-01

CONDITIONS: Group A β-Hemolytic Streptococci

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- oral and/or nasal specimen samples: After each patient has been tested according to conventional SOC and has enrolled in the study, up to ten oral and/or nasal specimen samples will be collected
  Interventions: Other: Collection of oral and/or nasal samples

INTERVENTIONS:
Other: Collection of oral and/or nasal samples — Collection of oral and/or nasal samples after SOC test performed

SUMMARY:
This prospective, sample collection study will assess different oral and/or nasal sample types collected from patients suspected of suffering from GABHS pharyngitis to conduct research and development on innovative GABHS detection methods specific for each sample type.

DETAILED DESCRIPTION:
Study candidates are patients age 3 and older with complaints of sore throat and are suspected of suffering from GABHS pharyngitis. Patients who consent and are found eligible will be enrolled in the study. Subjects will be tested according to the conventional standard of care in addition to providing extra specimen samples for the study.

After each patient has been tested according to conventional SOC and has enrolled in the study, up to ten oral and/or nasal specimen samples will be collected . Study participation is complete once all specimen samples are collected.

Most or all collected samples will be qualitatively tested and may also be quantitatively and/or semi-quantitatively tested for the presence of GABHS. Some collected samples may additionally or alternatively be tested for other respiratory infections as well. (such as SARS-CoV-2, influenza, etc.)

ELIGIBILITY:
Inclusion Criteria:

1. Patient, either male or female, is age 3 years or older;
2. Patient is suspected of suffering from GABHS pharyngitis, and is prescribed a throat culture by conventional SOC;
3. Patient or legal guardian is able to communicate with study personnel;
4. Patient or legal guardian is able to understand oral and written information regarding the nature of the study and is willing to provide written informed consent.

Exclusion Criteria:

1. Patients presently on antibiotics prescribed by a physician for treatment or prevention of GAS infection or has taken antibiotics within the past 3 days ( unless patient only first started taking antibiotics within the past 24 hour)
2. pregnancy
3. Patients who took mouth rinse or taking oral treatment for mouth sores within 3 hours of study

Min Age: 3 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The study population will be patients aged 3 years and older who are suspected of suffering from GABHS pharyngitis.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-11-18 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
quantify and compare the amount of GABHS | Study participation ( 1 day participation)
  quantify the amount of GABHS contained in different oral and/or nasal sample types collected from patients who have been diagnosed with GABHS pharyngitis
compare the amount of GABHS in different oral and/or nasal samlpes | Study participation ( 1 day participation)
  Compare the amount of GABHS contained in different oral and/or nasal sample types collected from patients who have been diagnosed with GABHS pharyngitis

SECONDARY OUTCOMES:
assess the efficacy of potential GABHS detection methods specifically designed for each oral and/or nasal sample type | Study participation ( 1 day participation)
  to assess the efficacy of potential GABHS detection methods specifically designed for each oral and/or nasal sample type by determining the sensitivity and specificity of each method in compare to the results from standard of care sampeling

CONTACTS AND LOCATIONS:
Locations (1):
- Leumit Healthcare services, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No